CLINICAL TRIAL: NCT05981560
Title: Effects of Closed Chain Exercise Versus Neuromuscular Training on Pain, Range of Motion, and Functional Performance in Football Players With Chronic Ankle Sprain
Brief Title: Effects of Closed Chain Exercise Versus Neuromuscular Training on Chronic Ankle Sprain in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0402
Record Dates: First submitted 2023-06-06; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Ankle Sprains; Chronic Pain
Keywords: Ankle Sprain; Chronic Ankle Instability; Exercise programs; Neuromuscular Training; Sports Injuries
MeSH Terms: conditions — Ankle Injuries; Chronic Pain; Athletic Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed Chain Exercise (Experimental): closed chain exercise plan given to the participant of this group
  Interventions: Other: Group A - Closed Chain Exercise
- Neuromuscular Training Exercise (Experimental): Neuromuscular training plan given to the participants of this group
  Interventions: Other: Group B - Neuromuscular Training Exercise

INTERVENTIONS:
Other: Group A - Closed Chain Exercise — 17 participants were in experimental group giving them closed chain exercise plan of 5 exercises, 10reps x 3sets each, on alternate 3 days per week for duration of 4-weeks, all values measured before and after 4-weeks
  Arms: Closed Chain Exercise
Other: Group B - Neuromuscular Training Exercise — 17 participants were in experimental group giving them neuromuscular training plan of 5 exercises, 10reps x 3sets each, on alternate 3 days per week for duration of 4-weeks, all values measured before and after 4-weeks.
  Arms: Neuromuscular Training Exercise

SUMMARY:
A current study will be conducted to determine the effects of closed-chain exercise versus neuromuscular training on pain, range of motion, and functional performance in football players with a chronic ankle sprain. This study will be a clinical trial conducted at the Pakistan sports board in the Lahore district. The study will be completed within the time duration of Six months. Non-probability convenient sampling technique will be used to collect the data. The sample size of 17 participants in each group will be taken in this study to find the effects of closed-chain exercise versus neuromuscular training on pain, range of motion, and functional performance in football players with a chronic ankle sprain. Athletes will be divided into two groups. Group A will be treated with closed-chain exercises and Group B will be with neuromuscular training. Pain (Numeric pain rating scale NPRS), Proprioceptive (balancing on a single leg with the eyes closed, balancing on a wobble board, Dynamic balance (Star Excursion Balance test and Y Balance Test), Functional Ankle Instability (Greek version of the Identification functional ankle instability questionnaire IdFAI), Cumberland Ankle Instability Tool (CHRONIC ANKLE INSTABILITY) and Ankle Instability Instrument (AII), Foot and Ankle Ability Measure (FAAM)-Sport Subscale, Range of Motion ROM (measure Goniometer) will be used as Data collecting tools. Three sessions of treatment per week for 4 weeks will be given. Data will be analyzed on SPSS version 22. In descriptive statistics Frequency tables, pie charts, and bar charts will be used to show the summary of group measurements measured over time.

DETAILED DESCRIPTION:
To determine the effects of closed-chain exercise versus neuromuscular training on pain, range of motion, and functional performance in football players with a chronic ankle sprain.

The study design will be a Randomized Clinical trial. Non-Probability Convenient Sampling will be used.

the sample size of 34 subjects is calculated.

TOOLS:

1. Pain (Numeric pain rating scale NPRS)
2. Range of Motion ROM (measure Goniometer)
3. Proprioceptive (balancing on a single leg with the eyes closed, balancing on a wobble board)
4. Dynamic balance (Star Excursion Balance test and Y Balance Test)
5. Functional Ankle Instability (Greek version of the Identification functional ankle instability questionnaire IdFAI)
6. Ankle Instability Instrument (AII)
7. Foot and Ankle Ability Measure (FAAM)-Sport Subscale The data will be analyzed using SPSS for Windows software, version 25. Statistical significance will be set at P= 0.05. After assessing the normality of the data by Shapiro wilk test it will be decided whether parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* • Both male and female

  * Age 18-35 (3)
  * Grade 1, 2 Ankle Sprain
  * Recurrent ankle Sprains (3)
  * Ankle Sprain Special Tests (Squeeze Test, Talar Tilt Test)

Exclusion Criteria:

* • Traumatic history or Ankle fracture (6 months)

  * any vestibular or balance disorders (1)
  * athletes who had suffered a sprain in the month prior to the start of the study(3)
  * who were taking anti-inflammatory drugs (3)
  * Poor physical fitness
  * Co-morbidities

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pain (NPRS Scale) | 4 weeks
  The Numeric Pain Rating Scale (NPRS) is a widely used tool for measuring and assessing pain intensity. It is a simple and subjective rating scale that allows individuals to quantify and communicate their level of pain on a numerical scale.
  The NPRS typically consists of a horizontal or vertical line with numbers ranging from 0 to 10. The numbers represent a continuum of pain intensity, where 0 represents "no pain" and 10 represents the "worst possible pain." The individual is asked to select the number that best corresponds to their current level of pain, with 0 indicating no pain and 10 indicating the most severe pain imaginable.
Range of Motion (Goniometer) | 4 weeks
  A goniometer is a measuring tool commonly used in healthcare and physical therapy to assess and quantify the range of motion (ROM) in joints. It consists of a stationary arm, a movable arm, and a protractor or scale to measure angles.
  To measure range of motion with a goniometer, the stationary arm is aligned with a fixed point on the body, typically an anatomical landmark associated with the joint being assessed. The movable arm is aligned with a second anatomical landmark, which moves as the joint is flexed or extended.
Functional Performance (Special Tests) | 4 weeks
  Functional performance refers to an individual's ability to perform everyday tasks and activities effectively and independently. It encompasses the physical, cognitive, and emotional skills required to carry out various activities that are necessary for daily living, work, leisure, and social participation.
  Functional performance is closely tied to an individual's overall functional capacity, which involves the integration of physical abilities, such as strength, endurance, balance, and coordination, with cognitive and emotional factors, including problem-solving, decision-making, attention, and motivation.
  The concept of functional performance extends beyond isolated movements or specific skills and focuses on how individuals function within their unique environments and roles.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alahmari KA, Kakaraparthi VN, Reddy RS, Silvian P, Tedla JS, Rengaramanujam K, Ahmad I. Combined Effects of Strengthening and Proprioceptive Training on Stability, Balance, and Proprioception Among Subjects with Chronic Ankle Instability in Different Age Groups: Evaluation of Clinical Outcome Measures. Indian J Orthop. 2020 Jul 15;55(Suppl 1):199-208. doi: 10.1007/s43465-020-00192-6. eCollection 2021 May. PMID 34122771
- [Background] Kachanathu S, Hafez A, Alenazi A, Hassan S, Algarni A, Albarrati AJPM, Rehabilitationsmedizin, Kurortmedizin. Efficacy of Closed and Open Kinematic Chain Exercises on Ankle Sprain Rehabilitation. 2016;26(01):28-31.
- [Background] Allois R, Niglia A, Pernice A, Cuesta-Barriuso R. Fascial therapy, strength exercises and taping in soccer players with recurrent ankle sprains: A randomized controlled trial. J Bodyw Mov Ther. 2021 Jul;27:256-264. doi: 10.1016/j.jbmt.2021.03.022. Epub 2021 Apr 2. PMID 34391242
- [Background] Shiravi Z, Shadmehr A, Moghadam ST, Moghadam BA. Comparison of dynamic postural stability scores between athletes with and without chronic ankle instability during lateral jump landing. Muscles Ligaments Tendons J. 2017 May 10;7(1):119-124. doi: 10.11138/mltj/2017.7.1.119. eCollection 2017 Jan-Mar. PMID 28717619
- [Background] Thompson JY, Byrne C, Williams MA, Keene DJ, Schlussel MM, Lamb SE. Prognostic factors for recovery following acute lateral ankle ligament sprain: a systematic review. BMC Musculoskelet Disord. 2017 Oct 23;18(1):421. doi: 10.1186/s12891-017-1777-9. PMID 29061135
- [Background] Greig M, McNaughton L. Soccer-specific fatigue decreases reactive postural control with implications for ankle sprain injury. Res Sports Med. 2014;22(4):368-79. doi: 10.1080/15438627.2014.944300. PMID 25295475
- [Background] Davenport TE, Kulig K, Fisher BE. Ankle manual therapy for individuals with post-acute ankle sprains: description of a randomized, placebo-controlled clinical trial. BMC Complement Altern Med. 2010 Oct 19;10:59. doi: 10.1186/1472-6882-10-59. PMID 20958995
- [Background] Czajka CM, Tran E, Cai AN, DiPreta JA. Ankle sprains and instability. Med Clin North Am. 2014 Mar;98(2):313-29. doi: 10.1016/j.mcna.2013.11.003. Epub 2014 Jan 10. PMID 24559877
- [Background] Faizullin I, Faizullina E. Effects of balance training on post-sprained ankle joint instability. Int J Risk Saf Med. 2015;27 Suppl 1:S99-S101. doi: 10.3233/JRS-150707. PMID 26639734
- [Background] Kim K, Jeon K. Development of an efficient rehabilitation exercise program for functional recovery in chronic ankle instability. J Phys Ther Sci. 2016 May;28(5):1443-7. doi: 10.1589/jpts.28.1443. Epub 2016 May 31. PMID 27313347
- [Background] McCall A, Carling C, Nedelec M, Davison M, Le Gall F, Berthoin S, Dupont G. Risk factors, testing and preventative strategies for non-contact injuries in professional football: current perceptions and practices of 44 teams from various premier leagues. Br J Sports Med. 2014 Sep;48(18):1352-7. doi: 10.1136/bjsports-2014-093439. Epub 2014 May 16. PMID 24837243
- [Background] Mohammadi Nia Samakosh H, Brito JP, Shojaedin SS, Hadadnezhad M, Oliveira R. What Does Provide Better Effects on Balance, Strength, and Lower Extremity Muscle Function in Professional Male Soccer Players with Chronic Ankle Instability? Hopping or a Balance Plus Strength Intervention? A Randomized Control Study. Healthcare (Basel). 2022 Sep 21;10(10):1822. doi: 10.3390/healthcare10101822. PMID 36292269
- [Background] Medina McKeon JM, Hoch MC. The Ankle-Joint Complex: A Kinesiologic Approach to Lateral Ankle Sprains. J Athl Train. 2019 Jun;54(6):589-602. doi: 10.4085/1062-6050-472-17. Epub 2019 Jun 11. PMID 31184957
- [Background] Hung YJ. Neuromuscular control and rehabilitation of the unstable ankle. World J Orthop. 2015 Jun 18;6(5):434-8. doi: 10.5312/wjo.v6.i5.434. eCollection 2015 Jun 18. PMID 26085985
- [Background] Owoeye OB, Akinbo SR, Tella BA, Olawale OA. Efficacy of the FIFA 11+ Warm-Up Programme in Male Youth Football: A Cluster Randomised Controlled Trial. J Sports Sci Med. 2014 May 1;13(2):321-8. eCollection 2014 May. PMID 24790486
- [Background] Emery CA, Roy TO, Whittaker JL, Nettel-Aguirre A, van Mechelen W. Neuromuscular training injury prevention strategies in youth sport: a systematic review and meta-analysis. Br J Sports Med. 2015 Jul;49(13):865-70. doi: 10.1136/bjsports-2015-094639. PMID 26084526
- [Background] Soomro N, Sanders R, Hackett D, Hubka T, Ebrahimi S, Freeston J, Cobley S. The Efficacy of Injury Prevention Programs in Adolescent Team Sports: A Meta-analysis. Am J Sports Med. 2016 Sep;44(9):2415-24. doi: 10.1177/0363546515618372. Epub 2015 Dec 16. PMID 26673035
- [Background] Owoeye OBA, Palacios-Derflingher LM, Emery CA. Prevention of Ankle Sprain Injuries in Youth Soccer and Basketball: Effectiveness of a Neuromuscular Training Program and Examining Risk Factors. Clin J Sport Med. 2018 Jul;28(4):325-331. doi: 10.1097/JSM.0000000000000462. PMID 29864071
- [Background] Caldemeyer LE, Brown SM, Mulcahey MK. Neuromuscular training for the prevention of ankle sprains in female athletes: a systematic review. Phys Sportsmed. 2020 Nov;48(4):363-369. doi: 10.1080/00913847.2020.1732246. Epub 2020 Feb 28. PMID 32067546
- [Background] Kaminski TW, Hertel J, Amendola N, Docherty CL, Dolan MG, Hopkins JT, Nussbaum E, Poppy W, Richie D; National Athletic Trainers' Association. National Athletic Trainers' Association position statement: conservative management and prevention of ankle sprains in athletes. J Athl Train. 2013 Jul-Aug;48(4):528-45. doi: 10.4085/1062-6050-48.4.02. PMID 23855363
- [Background] O'Driscoll J, Delahunt E. Neuromuscular training to enhance sensorimotor and functional deficits in subjects with chronic ankle instability: A systematic review and best evidence synthesis. Sports Med Arthrosc Rehabil Ther Technol. 2011 Sep 22;3:19. doi: 10.1186/1758-2555-3-19. PMID 21939557